CLINICAL TRIAL: NCT02348463
Title: Treatment of Bacterial Vaginosis in Early Pregnancy in Skaraborg County in Sweden and the Effect on Spontaneous Preterm Delivery
Brief Title: Treatment of Bacterial Vaginosis in Early Pregnancy in Skaraborg and the Effect on Spontaneous Preterm Delivery
Status: Completed | Type: Observational
Sponsor: Skaraborg Hospital (Other Government)
Responsible Party: Principal Investigator, Per-Goran Larsson, Professor Consultat, Skaraborg Hospital
Other Study IDs: BV and pregnancy
Record Dates: First submitted 2014-11-28; First posted 2015-01-28 (Estimated); Last update posted 2015-01-28 (Estimated); Status verified 2015-01

CONDITIONS: Bacterial Vaginosis
MeSH Terms: conditions — Vaginosis, Bacterial | interventions — clindamycin phosphate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- treatment of bacterial vaginosis: women with bacterial vaginosis will be offered treatment with clindamycin-2-phosphate
  Interventions: Drug: Clindamycin-2-phosphate

INTERVENTIONS:
Drug: Clindamycin-2-phosphate — how many women will deliver before the 37th week of gestation
  Other Names: Dalacin vaginal cream

SUMMARY:
Bacterial vaginosis (BV) is a known risk factor for preterm delivery. This study was conducted in an attempt to investigate if treatment of bacterial vaginosis in early pregnancy could reduce the risk for preterm delivery.

Women were screened for bacterial vaginosis during the first visits at the maternal health care unit with a vaginal sample that were taken by the midwife or by herself. After the vaginal samples was air dried it was sent to the gynaecological department and was investigated using Hay/Ison classification. Eligible women were those who had lived in Skaraborg and delivered at Skaraborg hospital.

DETAILED DESCRIPTION:
The study has started 2007 and will continue until 2014. Pregnant women that will come to the maternal health care units in gestational week 8-11 will be offered to be screened for bacterial vaginosis. A vaginal sample will be taken by the midwife or by the women herself. The vaginal sample is air-dried and sent to the gynecological. There it is investigated using Hay/Ison classification for the diagnosis of bacterial vaginosis.

Women with bacterial vaginosis will be offered treatment with topical clindamycin treatment for 7 days if the women has passed the 12th gestational week. A control sample for the test of cure will be done after 10 week. If not cured of BV she will be offered a new treatment.

All women will be followed until delivery.

ELIGIBILITY:
Inclusion Criteria:

* pregnant women screened for bacterial vaginosis in early pregnancy

Exclusion Criteria:

* women not delivered at Skaraborg hospital.

Ages: 18 Years to 52 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Pregnant women with bacterial vaginosis in early pregnancy
Sampling Method: Probability Sample
Enrollment: 540 (Actual)
Dates: Start 2007-01; Primary Completion 2013-12 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
preterm delivery | before 37th week of gestation

SECONDARY OUTCOMES:
cure of bacterial vaginosis | after 10 weeks